CLINICAL TRIAL: NCT06068504
Title: Shear Stress in the Arteries of the Lower Limbs During Arm Cranking Exercise in Patients With Peripheral Arterial Disease
Brief Title: Shear Stress in the Arteries of the Lower Limbs During Exercise in Patients With Peripheral Arterial Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Raphael Mendes Ritti Dias, Principal Investigator, University of Nove de Julho
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Heating_PAD
Record Dates: First submitted 2023-09-22; First posted 2023-10-05 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Peripheral Arterial Disease
Keywords: exercise; arm-cranking; vascular function
MeSH Terms: conditions — Peripheral Arterial Disease; Motor Activity | interventions — Exercise Test; Exercise; Heating

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm-cranking exercise (Experimental): Patients will be perform arm-cranking exercise. The exercise will be performed in 15 sets of 2 min of exercise at a moderate intensity (13-15 in Borg scale)
  Interventions: Other: Arm-cranking exercise
- Heating (Active Comparator): Patients will perform 15 sets of 2 min of immersion of their foot in a warm water (42 degrees)
  Interventions: Other: Heating
- Control (No Intervention): Patients will remain seated for 60 min

INTERVENTIONS:
Other: Arm-cranking exercise — Arm-cranking exercise
  Other Names: Arm exercise; Exercise
  Arms: Arm-cranking exercise
Other: Heating — Immersion of the foot in warm water
  Arms: Heating

SUMMARY:
The aim of the study will be to evaluate shear stress and blood flow parameters in lower limb arteries during arm cycle ergometer exercise in participants with peripheral artery disease. Twenty patients participants with peripheral artery disease and claudication symptoms will be recruited. Participants will perform 3 experimental sessions in random order. Iarm-cranking (15 sets of two minutes exercise), warm water foot immersion, and control. During the interventions, blood pressure and heart rate will be assessed every 6 minutes. Measurements of arterial diameter, blood flow, anterograde and retrograde shear stress of the femoral artery will be evaluated using a two-dimensional ultrasound device with spectral Doppler.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of peripheral artery disease or ankle-brachial index less than 0.90 in one or both limbs
* do not present peripheral neuropathy;
* be able to exercise after medical approval
* aged 50 or over.

Exclusion Criteria:

* Medication change during the study
* Health problems that contraindicates the practice of physical exercise.

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Femoral artery diameter [mm] | Before the intervention and at 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 28, and 30 minutes into the intervention
  Measurements will be obtained through duplex ultrasound in accordance with global recommendations.
Femoral artery shear rate [sec.-1] | Before the intervention and at 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 28, and 30 minutes into the intervention
  Measurements will be obtained through duplex ultrasound in accordance with global recommendations.
Femoral artery Blood flow [mL/min] | Before the intervention and at 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 28, and 30 minutes into the intervention
  Measurements will be obtained through duplex ultrasound in accordance with global recommendations.

SECONDARY OUTCOMES:
Brachial systolic and diastolic blood pressure [mmHg] | Before the intervention and at 1, 3, 5, 7, 9, 11, 13, 15, 17, 19, 21, 23, 25, 27, and 29 minutes into the intervention
  Systolic and diastolic blood pressures will be assessment in the arms with an automatic blood pressure monitor (HEM-742, Omron Healthcare, Japan)
Heart rate [bpm] | Before and up to 30 minutes into the intervention
  Heart rate assessment with a heart rate monitor (Polar H10, Polar®, Finland)

CONTACTS AND LOCATIONS:
Overall Officials: Raphael Dias, Principal Investigator — University of Nove de Julho
Locations (1):
- University Nove de Julho, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: One year after the study completion
Access Criteria: Upon request